CLINICAL TRIAL: NCT03565185
Title: Comparison Of An Exoskeleton Device With An End-Effector Device In Robotic Gait Assesment Of Stroke
Brief Title: Comparison Of Two Different Type Robot Assisted Gait Training In Rehabilitation Of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erenköy Physical Therapy and Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, AYLİN SARI, Medical Doctor,, Erenköy Physical Therapy and Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ErenkoyPTRH
Record Dates: First submitted 2018-05-21; First posted 2018-06-21 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- End-effector (Active Comparator): For stroke rehabilitation 5 days a week in addition to conventional treatment methods robot-assisted gait training(end-effector type-Lokohelp) will be taken with 45 minutes a day for 3 days a week for 4 weeks.
  Patients will be assessed with PASS, Rivermead mobility index, 10-meter walking test, 6-minute walking test, Barthel index, and FAC in terms of baseline and ending for posture, mobility, walking velocity, walking capacity, daily life activities and ambulance level.
  Interventions: Other: robot-assisted gait training
- Exoskeleton (Active Comparator): For stroke rehabilitation 5 days a week in addition to conventional treatment methods robot-assisted gait training (exoskeleton type-Robogait) will be taken with 45 minutes a day for 3 days a week for 4 weeks.
  Patients will be assessed with PASS, Rivermead mobility index, 10-meter walking test, 6-minute walking test, Barthel index, and FAC in terms of baseline and ending for posture, mobility, walking velocity, walking capacity, daily life activities and ambulance level.
  Interventions: Other: robot-assisted gait training
- conventional treatment (Placebo Comparator): conventional treatment methods for stroke rehabilitation 5 days a week Patients will be assessed with PASS, Rivermead mobility index, 10-meter walking test, 6-minute walking test, Barthel index, and FAC in terms of baseline and ending for posture, mobility, walking velocity, walking capacity, daily life activities and ambulance level.
  Interventions: Other: placebo

INTERVENTIONS:
Other: robot-assisted gait training — Investigators will use robot-assisted gait training for rehabilitation of stroke
  Arms: End-effector; Exoskeleton
Other: placebo — Investigators will use only conventional treatment without robot-assisted gait training
  Other Names: conventional treatment
  Arms: conventional treatment

SUMMARY:
Investigators aimed to compare the results of rehabilitation with an exoskeleton device(Robogait) and with an end-effector device(Lokohelp)

DETAILED DESCRIPTION:
There are different types of devices in robotic rehabilitation which has been used in recent years for stroke. Investigators aimed to compare the results of rehabilitation with an exoskeleton device(Robogait) and with an end-effector device(Lokohelp) in robot-assisted gait training of stroke rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Rehabilitation need for stroke
* Patients under FAC stage 4
* No contraindications for robotic rehabilitation
* Subacute stroke

Exclusion Criteria:

* The robot-orthosis does not fit the patient's body
* Inadequate body weight (obesity)
* Severe contractures
* Bone instability (nonstable spinal cord fracture and severe osteoporosis)
* Circulation problems
* Cardiac problems
* Open wounds on the lower extremities or in the body where they will come into contact with the orthosis
* Uncoordinated, psychotic or aggressive patients
* Serious cognitive disorders
* Patients with long-term infusion therapy
* Hip, knee, ankle arthrodesis
* Epilepsy
* Patients with disproportionate limb or vertebrae, such as bone cartilage dysplasia
* Those with severe vascular problems of the lower extremity
* Conditions requiring rest or immobilization, such as osteomyelitis and other inflammatory/infectious diseases
* Severe respiratory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | 4 weeks
  6 minute walk test for walking speed
10 meter walking test | 4 weeks
  10 meter walking test for walking
Postural Assessment Scale for Stroke(PASS) | 4 weeks
  Postural Assessment Scale for Stroke(PASS) will be used

SECONDARY OUTCOMES:
FAC(Functional Ambulation Classification) | 4 weeks
  FAC will be used for ambulation
Barthel Index | 4 weeks
  Barthel Index will be used for daily living activities

CONTACTS AND LOCATIONS:
Overall Officials: Aylin SARI, Study Chair — Dr.
Locations (1):
- Erenkoy physical treatment and rehabilitation hospital, Istanbul, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No